CLINICAL TRIAL: NCT00185900
Title: Magnesium Sulfate Versus Nifedipine for the Acute Tocolysis of Preterm Labor: A Prospective, Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76145
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-10

CONDITIONS: Obstetric Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Magnesium Sulfate; Nifedipine

ARMS (2):
- Magnesium Sulfate (Active Comparator): Preterm labor treatment with Magnesium Sulfate.
  Interventions: Drug: Magnesium Sulfate
- Nifedipine (Active Comparator): Preterm labor treatment with Nifedipine.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Magnesium Sulfate — Preterm labor treatment with Magnesium Sulfate 4 gram bolus followed by 2 gm per hour infusion. 2 Gm bolus as needed and/or rate increase up to 4gm per hour were allowed at the discretion of the treating physician.
  Arms: Magnesium Sulfate
Drug: Nifedipine — Preterm labor treatment with Nifedipine 10 mg. sublingually every 20 minutes for three doses, followed by 20 mg. orally every 4 or 6 hours.
  Arms: Nifedipine

SUMMARY:
To compare intravenous magnesium sulfate to oral nifedipine for acute tocolysis of preterm labor

ELIGIBILITY:
Inclusion Criteria::- Uterine contractions and cervical change or ruptured membranes in a preterm gestation Exclusion Criteria:- placental abruption, fetal distress, placenta previa, maternal medical contraindication to tocolysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 1999-04; Primary Completion 2005-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lyell DJ, Pullen K, Campbell L, Ching S, Druzin ML, Chitkara U, Burrs D, Caughey AB, El-Sayed YY. Magnesium sulfate compared with nifedipine for acute tocolysis of preterm labor: a randomized controlled trial. Obstet Gynecol. 2007 Jul;110(1):61-7. doi: 10.1097/01.AOG.0000269048.06634.35. PMID 17601897
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- See also: Obstet Gynecol. 2007 Jul;110(1):61-7. — http://www.greenjournal.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnesium Sulfate | Nifedipine
Started | 92 | 100
Completed | 92 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulfate | Nifedipine | Total
Number analyzed (Participants) | 92 | 100 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (6.8) | 26.3 (6.3) | 26.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 100 | 192
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 92 | 100 | 192

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prevention of Preterm Delivery for 48 Hours With Attainment of Uterine Quiescence
Description: Uterine quiescence defined by 12 hours of six or fewer contractions per hour and no further cervical change within 48 hours of tocolytic initiation.
Time Frame: 48 hours after administration of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulfate | Nifedipine
Number analyzed (Participants) | 92 | 100
Participants | 80 | 72
Statistical Analysis 1: Comparison: Magnesium Sulfate vs Nifedipine; Test type: Superiority; p = 0.01, Chi-squared

2. Secondary Outcome: Time to Uterine Quiescence
Description: Uterine quiescence was defined by 12 hours of six of fewer contractions per hour and no further cervical change.
Time Frame: Until delivery, up to 42 weeks of gestation
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Magnesium Sulfate | Nifedipine
Number analyzed (Participants) | 92 | 100
hours | 8.4 (6.5) | 6.1 (6.3)

3. Secondary Outcome: Gestational Age at Delivery
Description: Presented as weeks
Time Frame: Until delivery, up to 42 weeks of gestation
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Magnesium Sulfate | Nifedipine
Number analyzed (Participants) | 92 | 100
weeks | 35.8 (3.4) | 36.0 (3.1)

4. Secondary Outcome: Neonatal Birth Weight
Description: Presented as grams
Time Frame: Until delivery, up to 42 weeks of gestation
Population: Data included twins, so the group totals are greater than seen in the Overall Number of Participants Analyzed
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Magnesium Sulfate | Nifedipine
Number analyzed (Participants) | 106 | 110
grams | 2550 (802) | 2650 (698)

5. Secondary Outcome: Serious Maternal Adverse Effect
Description: A composite of any of the following: chest pain, pulmonary edema, shortness of breath or hypotension.
Time Frame: From study enrollment until discharge from delivery hospital, up to 30 days after delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulfate | Nifedipine
Number analyzed (Participants) | 92 | 100
Participants | 20 | 10

6. Secondary Outcome: Composite Neonatal Morbidity
Description: Defined as any of the following: respiratory distress syndrome, intraventricular hemorrhage, necrotizing enterocolitis, sepsis or fetal/neonatal death.
Time Frame: From delivery until discharge from the hospital, up to 30 days of age
Population: Data included twins, so the group totals are greater than seen in the Overall Number of Participants Analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium Sulfate | Nifedipine
Number analyzed (Participants) | 106 | 110
Participants | 27 | 22

ADVERSE EVENTS:
Time Frame: From study enrollment until discharge from the delivery hospital, up to 30 days after delivery.
Description: Adverse events were assessed by patient interview from a list of adverse effects and chart review.
Arm/Group | Magnesium Sulfate | Nifedipine
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/100
Serious Adverse Events (participants affected / at risk) | 25/92 | 12/100
Other Adverse Events (participants affected / at risk) | 29/92 | 22/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magnesium Sulfate (N=92) | Nifedipine (N=100)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 3
Chest pain (Cardiac disorders) | 7 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magnesium Sulfate (N=92) | Nifedipine (N=100)
Nausea (Gastrointestinal disorders) | 29 | 6
Lethargy (Nervous system disorders) | 27 | 3
Vomiting (Gastrointestinal disorders) | 24 | 5
Flushing (Skin and subcutaneous tissue disorders) | 20 | 1
Blurry Vision (Eye disorders) | 12 | 0
Dizziness (Nervous system disorders) | 16 | 3
Double vision (Eye disorders) | 3 | 0
Headache (Nervous system disorders) | 11 | 22
Palpitations (Cardiac disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No